CLINICAL TRIAL: NCT02554825
Title: Healthy Futures Longitudinal School-Cluster Randomized Controlled Trial
Brief Title: Healthy Futures Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JSI Research & Training Institute, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Black Ministerial Alliance of Greater Boston (Other); Healthy Futures (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: JSI R&T #13-012
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Sexual Behavior
MeSH Terms: conditions — Sexual Behavior

ARMS (2):
- Healthy Futures (Experimental)
  Interventions: Behavioral: Healthy Futures
- Control (Other)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Healthy Futures — Healthy Futures is an age-appropriate program that targets change at different social ecological levels-individual, interpersonal, and organizational. The main component is a classroom-based relationship education curriculum, Nu-CULTURE, offered in 6th, 7th, and 8th grade for eight 50-minute sessions each year. A number of supplemental efforts aim to enhance the Nu-CULTURE program and create social supports: 1) virtual classrooms where participating youth are encouraged to visit age-appropriate youth websites; 2) daily interactive parental connection forms linked with Nu-CULTURE, a parent website, and workshops (True Connections); 3) a 10-week after-school program, Rhymin' it Write, encourages youth leadership; 4) a 6-week summer program, Code A, engages youth during out-of-school time after 8th grade.
  Arms: Healthy Futures
Behavioral: Control — The Control Curriculum offers students in the control group two 50-minute classes each year on general health education topics. Students in the 6th grade receive a class on puberty/reproduction and a class on bullying prevention; students in the 7th grade receive two classes on dating-violence prevention; and students in the 8th grade receive two classes on mental health promotion.
  Arms: Control

SUMMARY:
This study evaluated the impact of the three-year Healthy Futures program on teen sexual behaviors in three Massachusetts cities.

DETAILED DESCRIPTION:
This study evaluated the impact of the three-year Healthy Futures program on teen sexual behaviors in three Massachusetts cities. This longitudinal school-cluster randomized controlled trial included 15 public middle schools (n=1,344). Participants were enrolled in the 6th grade in the 2011-2012 school year (Cohort 1) or 2012-2013 school year (Cohort 2). Outcome data sources included five student surveys: baseline; 6th, 7th, 8th grade follow-ups; and 9th grade follow-up (Cohort 1 only).

ELIGIBILITY:
Inclusion Criteria:

* Students attended one of the 15 participating public middle schools
* Students were enrolled in the 6th grade in the 2011-2012 school year (Cohort 1) or 2012-2013 school year (Cohort 2)
* Students were not withdrawn from Healthy Futures program participation by himself/herself, a parent, or school administrator(s) prior to the consent/assent process for the study

Exclusion Criteria:

* Students were were not in the 6th grade at the time of consent
* Students were not in the school after the consent/assent process occurred
* Students were withdrawn from Healthy Futures program participation by himself/herself, a parent, or school administrator(s) prior to the consent/assent process for the study.

Ages: 10 Years to 15 Years | Sex: All
Age Groups: Child
Enrollment: 1344 (Actual)
Dates: Start 2011-08; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of participants who reported vaginal sex | 2 Years
  Participants were followed for the duration of the three-year Healthy Futures program delivered in 6th, 7th, and 8th grades. The primary outcome was measured approximately two years (8th grade) after the baseline (6th grade) questionnaire.
  Prevalence of participants who reported vaginal sex was measured by participant response [Yes/No] to the question: "For the purposes of this survey, by sex, we mean a male putting his penis into a female's vagina. Other ways of saying sex are "doing it" or going all the way". Have you ever had sex?"

CONTACTS AND LOCATIONS:
Locations (1):
- JSI Research & Training Institute, Inc., Boston, Massachusetts, United States